CLINICAL TRIAL: NCT01356602
Title: A Randomized, Double-blind, Active-controlled Study of Canakinumab Prefilled Syringes or Reconstituted Lyophilizate Versus Triamcinolone Acetonide for Treating Acute Gouty Arthritis Flares in Frequently Flaring Patients
Brief Title: Safety and Efficacy of Canakinumab Prefilled Syringes in Frequently Flaring Acute Gouty Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885H2361; 2010-024173-39 (EudraCT Number)
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Acute Gouty Arthritis
Keywords: Gout; arthritis; gout flare; acute gout; gouty; rheumatic disease; uric acid
MeSH Terms: conditions — Gout; Arthritis; Rheumatic Diseases | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Canakinumab, pre-filled syringes (PFS) (Experimental): Patients on this arm received 150 mg subcutaneously (s.c.) at randomization and upon new flare. The doses were provided as pre-filled syringes. The patients were given 3 injections: two placebo and one active drug.
  Interventions: Drug: Canakinumab pre-filled syringe; Drug: Placebo
- Canakinumab, lyophilizate (LYO) (Active Comparator): The patients on this arm received 150 mg s.c. at randomization and upon new flare. The doses were provided as lyophilized powder and had to be reconstituted with water for injection before application. The patients were given 3 injections: two placebo and one active drug.
  Interventions: Drug: Canakinumab lyophilized powder; Drug: Placebo
- Triamcinolone Acetonide (Active Comparator): The patients on this arm received 40 mg intramuscular (i.m.) at randomization and upon new flare. The patients were given 3 injections: two placebo and one active drug.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab pre-filled syringe — Canakinumab pre-filled syringe
  Arms: Canakinumab, pre-filled syringes (PFS)
Drug: Canakinumab lyophilized powder — Canakinumab lyophilized powder
  Arms: Canakinumab, lyophilizate (LYO)
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide
  Arms: Triamcinolone Acetonide
Drug: Placebo — Matching placebo to Canakinumab (PFS), Canakinumab (LYO) and Triamcinolone Acetonide

SUMMARY:
This study assessed the safety and efficacy of canakinumab pre-filled syringes in comparison to triamcinolone acetonide 40 mg and canakinumab lyophilizate in patients that have frequent flares of acute gouty arthritis.

ELIGIBILITY:
Inclusion criteria:

* 3 or more gout flares within last year
* Contraindication, intolerance or lack of efficacy for NSAIDs and/or colchicine
* Body mass index of less than or equal to 45 kg/m2

Exclusion criteria:

* Use of the following therapies (within varying protocol defined timeframes): corticosteroids, narcotics, topical ice/cold packs, chronic opiate treatment, NSAIDs (such as aspirin), colchicine.
* Hemodialysis
* Live vaccine within 3 months before first dose
* Donation or loss of 400 mL or more within 3 months before first dose
* Gout brought on by other factors such as chemotherapy, lead, transplant, etc.
* Presence of other acute inflammatory arthritis such as Rheumatoid Arthritis
* Any conditions or significant medical problems that puts the patient at an unacceptable immunological risk to receive this type of therapy such as HIV, Hepatitis, Tuberculosis and other infections/conditions
* Significant cardiovascular conditions such as uncontrolled hypertension
* Significant medical diseases such as uncontrolled diabetes, thyroid disease
* History of malignancy of any organ system within the past 5 years
* Women who are pregnant or nursing
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (91):
- United States (65):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Gulf Shores, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Fair Oaks, California
  - Novartis Investigative Site, Norwalk, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Westlake Village, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Meridian, Idaho
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, Roslyn, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Mogadore, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Murrells Inlet, South Carolina
  - Novartis Investigative Site, Ninety Six, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Bristol, Tennessee
  - Novartis Investigative Site, Fayetteville, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Bellevue, Washington
- Canada (4):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Germany (9):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Messkirch
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Weener
  - Novartis Investigative Site, Zwiesel
- Hungary (9):
  - Novartis Investigative Site, Szikszó, Hungary
  - Novartis Investigative Site, Békéscsaba
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Veszprém
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of subjects randomized was 397. Only 389 subjects (including one subject with 3 placebo injections) received study drug (Safety set). Subjects who received more than one active dose were counted in each treatment group, leading to a safety set of 399 subjects. Subjects who did not receive study drug were excluded from analysis.
Groups:
- Canakinumab, Lyophilizate (LYO): The patients on this arm received 150 mg s.c. at randomization and upon new flare. The doses were provided as lyophilized power and had to be reconstituted with water for injection before application. The patients were given 3 injections: two placebo and one active drug.
Period: Overall Study
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Started | 133 | 132 | 132
Safety Set | 133 (In this arm, 1 patient had only 3 placebo injections and 3 patients also took other active drug.) | 133 (In this arm, 3 patients also took other active drug.) | 133 (In this arm, 3 patients also took other active drug.)
Full Analysis Set | 131 | 129 | 129
Completed | 124 | 117 | 108
Not Completed | 9 | 15 | 24
Not completed — Protocol Deviation | 0 | 1 | 1
Not completed — Administrative Problems | 1 | 4 | 5
Not completed — Lost to Follow-up | 4 | 5 | 6
Not completed — Withdrawal by Subject | 4 | 3 | 7
Not completed — Lack of Efficacy | 0 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide | Total
Number analyzed (Participants) | 133 | 133 | 133 | 399
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (11.21) | 53 (11.84) | 53.7 (11.33) | 53.5 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 11 | 35
  Male | 118 | 124 | 122 | 364

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity on a 0-100 mm Visual Analog Scale (VAS) Between the Canakinumab 150 mg PFS and Triamcinolone Acetonide 40 mg Groups
Description: The Visual Analog Scale (VAS) is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. The VAS contains a continuous line between two end points whereby the respondent places a mark on the line to indicate his or her response. In this study, patients scored their pain intensity in the most affected joint of the gout flare on a 0 100 mm VAS. The scale ranged from 0 (no pain) to 100 (unbearable pain). The scores were measured to the nearest millimeter from the left. Missing pain intensity data at 72 hours was imputed using the Last-Observation-Carried-Forward (LOCF) method.
Time Frame: 72 hours post dose
Population: Full Analysis Set: The Full Analysis Set (FAS) consisted of all patients as randomized that had at least one dose of study drug. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: Millimeters
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 130 | 0 | 126
Millimeters | 17.1 (2.04) |  | 32 (2.08)

2. Secondary Outcome: Pain Intensity on a 0 - 100 mm VAS Between the Canakinumab 150 mg PFS and Canakinumab 150 mg LYO Groups
Description: as for outcome 1
Time Frame: 72 hours post dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimeters
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 130 | 129 | 0
Millimeters | 17.1 (2.04) | 19.7 (2.05) |

3. Secondary Outcome: Patient's Assessment of Pain Intensity on a 0-100mm VAS
Description: The Visual Analog Scale (VAS) is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. The VAS contains a continuous line between two end points whereby the respondent places a mark on the line to indicate his or her response. In this study, patients scored their pain intensity in the most affected joint of the gout flare on a 0 100 mm VAS. The scale ranged from 0 (no pain) to 100 (unbearable pain). The scores were measured to the nearest millimeter from the left. The LOCF method was used to impute post-dose pain intensity VAS measurements up to 14 days.
Time Frame: 14 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimeters
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 130 | 129 | 126
Millimeters | 7.9 (1.69) | 8.2 (1.7) | 14.8 (1.72)

4. Secondary Outcome: Patient's Assessment of Pain Intensity on a 5-point Likert Scale
Description: A Likert scale is a type of scale with a range of responses corresponding to an item such as pain. The respondent selects the best response that indicates the respondent's subjective evaluation of the item. Patients scored their pain intensity in the most affected joint of the gout flare on a 5-point Likert scale (none, mild, moderate, severe, extreme). The scores were measured to the nearest millimeter from the left. The LOCF method was used to impute post-dose pain intensity Likert measurements up to 14 days.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 128
Percentage of Patients
  None | 35.9 | 32.6 | 23.4
  Mild | 45.8 | 44.2 | 36.7
  Moderate | 15.3 | 21.7 | 21.9
  Severe | 2.3 | 1.6 | 14.1
  Extreme | 0.8 | 0 | 3.9

5. Secondary Outcome: Number of Patients With at Least One New Gouty Arthritis Flare After Baseline
Description: Patients met the definition of a new flare if they had: a flare in a joint, which was not a previously affected joint (at baseline or during the study), or a flare in a joint previously affected (at baseline or during the study) after the previous flare in that joint had resolved completely according to the patient's perception. Patients did NOT meet the criterion of having a new gout flare if they had increasing/renewed gout pain in an affected joint before the flare had resolved completely.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Particpants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Particpants | 12 | 12 | 52

6. Secondary Outcome: Time to the First New Gouty Arthritis Flare
Description: Patients met the definition of a new flare if they had: a flare in a joint, which was not a previously affected joint (at baseline or during the study), or a flare in a joint previously affected (at baseline or during the study) after the previous flare in that joint had resolved completely according to the patient's perception. Patients did NOT meet the criterion of having a new gout flare if they had increasing/renewed gout pain in an affected joint before the flare had resolved completely. Less than 50% of patients had new flares. Therefore, the median time to new flare could not be calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Days | NA [NA to NA] — Less than 50% of patients had new flares. Therefore, the median time to new flare could not be calculated. | NA [NA to NA] — Less than 50% of patients had new flares. Therefore, the median time to new flare could not be calculated. | NA [NA to NA] — Less than 50% of patients had new flares. Therefore, the median time to new flare could not be calculated.

7. Secondary Outcome: Time to 50% Reduction in Baseline Pain on a 0 - 100 VAS
Description: The Visual Analog Scale (VAS) is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. The VAS contains a continuous line between two end points whereby the respondent places a mark on the line to indicate his or her response. In this study, patients scored their pain intensity in the most affected joint of the gout flare on a 0 100 mm VAS. The scale ranged from 0 (no pain) to 100 (unbearable pain). The scores were measured to the nearest millimeter from the left. Kaplan Meier estimate of time to 50% reduction in baseline pain, along with associated 95% confidence interval, were reported.
Time Frame: 14 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 130 | 129 | 129
Hours | 24 [22 to 25] | 25 [24 to 48] | 48 [25 to 54]

8. Secondary Outcome: Time to Resolution of Gouty Arthritis Flare as Reported by Patient
Description: Patients completed diary entries at 6, 12, 24, 48 and 72 hours post dose and then daily up to 7 days post-dose and/or daily until resolution of the flare. Kaplan Meier estimate of time to resolution of gouty flare as reported by patient, along with associated 95% confiedence interval, were reported.
Time Frame: 14 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 128 | 129
Hours | 142 [96 to 168] | 120 [96 to 145] | 170 [144 to 216]

9. Secondary Outcome: Patient's Global Assessment of Response to Treatment on a 5-point Likert Scale
Description: A Likert scale is a type of scale with a range of responses corresponding to an item such as pain. The respondent selects the best response that indicates the respondent's subjective evaluation of the item. Patients scored their response to treatment on a 5-point Likert scale (excellent, good, acceptable, slight, poor). This outcome measure shows the number of patients indicating each score on the scale.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Participants
  Excellent | 36.0 | 34.8 | 20.4
  Good | 43.2 | 36.5 | 31.9
  Acceptable | 10.4 | 20.0 | 21.2
  Slight | 6.4 | 7.8 | 14.2
  Poor | 4.0 | 0.9 | 12.4

10. Secondary Outcome: Physician's Global Assessment of Response to Treatment on a 5 Point Likert Scale
Description: A Likert scale is a type of scale with a range of responses corresponding to an item such as pain. The respondent selects the best response that indicates the respondent's subjective evaluation of the item. Study physicians scored their assessment of the patients' response to treatment on a 5-point Likert scale (very good, good, fair, poor, very poor).
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Participants
  Very good | 46.2 | 33.6 | 21.5
  Good | 35.4 | 48.8 | 33.9
  Fair | 15.4 | 16.0 | 23.1
  Poor | 1.5 | 1.6 | 14.0
  Very poor | 1.5 | 0.0 | 7.4

11. Secondary Outcome: Physician's Assessment of Tenderness
Description: The study physician assessed the most affected joint for tenderness. Tenderness was measured on a 0 - 3 point scale as follows: 0 = no pain, 1 = patient states that "there is pain", 2 = patient states "there is pain and winces" and 3 = patient states "there is pain, winces and withdraws" on palpation or passive movement of the affected study joint.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Participants
  No pain | 50.0 | 40.0 | 29.8
  There is pain | 43.1 | 52.8 | 47.1
  There is pain and winces | 5.4 | 6.4 | 14.0
  There is pain, winces and withdraws | 1.5 | 0.8 | 9.1

12. Secondary Outcome: Physician's Assessment of Swelling
Description: The study physician assessed the most affected joint for swelling. Swelling was measured on a 0 - 3 point scale as follows: 0 = no swelling, 1 = palpable, 2= visible and 3 = bulging beyond the joint margins.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Partipants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Partipants
  No swelling | 60.8 | 55.2 | 51.2
  Palpable | 26.9 | 25.6 | 15.7
  Visible | 10.8 | 17.6 | 24.8
  Bulging beyond the joint margins | 1.5 | 1.6 | 8.3

13. Secondary Outcome: Physician's Assessment of Erythema
Description: The study physician assessed the most affected joint for erythema. Erythema was assessed as present, absent or not assessable.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Participants
  Absent | 88.3 | 82.9 | 68.6
  Present | 11.7 | 17.1 | 31.4

14. Secondary Outcome: Physician's Assessment of Range of Motion of the Most Affected Joint
Description: The study physician assessed the patient's range of motion of the most affected joint on a 5 point Likert scale (normal, mildly restricted, moderately restricted, severely restricted and immobilized).
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Participants
  Normal | 50.0 | 44.8 | 35.5
  Mildly restricted | 37.7 | 40.8 | 37.2
  Moderately restricted | 11.5 | 12.0 | 14.0
  Severely restricted | 0.8 | 2.4 | 12.4
  Immobilized | 0.0 | 0.0 | 0.8

15. Secondary Outcome: Proportion of Patients With Rescue Medication Intake
Description: Patients used a diary to record the time of intake of rescue medication and the amount taken.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Particpants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Percentage of Particpants | 29.0 | 31.8 | 45.7

16. Secondary Outcome: Time to First Rescue Medication Intake
Description: Patients used a diary to record the time of intake of rescue medication and the amount taken.
Time Frame: 14 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 38 | 40 | 59
Hours | 11 (61.87) [4 to 279] | 7.5 (31.59) [3 to 142] | 11 (39.06) [1 to 186]

17. Secondary Outcome: Amount of Rescue Medication Taken (mg)
Description: Patients used a diary to record the time of intake of rescue medication and the amount taken.
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
milligrams (mg)
  Acetaminophen | 609.2 (1800.06) | 1108.3 (2821.54) | 2323.1 (5580.82)
  Codeine | 12.7 (55.30) | 23.9 (124.56) | 60.8 (191.2)
  Prednisolone / Prednisone | 5.8 (23.13) | 6.7 (25.09) | 24.7 (53.20)

18. Secondary Outcome: C-reactive Protein Level
Description: A central laboratory was used for analysis of all blood samples collected.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg / L
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 123 | 119 | 118
mg / L | 3.65 [3.11 to 4.29] | 3.37 [2.86 to 3.96] | 5.2 [4.41 to 6.13]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Only 389 subjects (including one subject with 3 placebo injections) received study drug (Safety set). Subjects who received more than one active dose were counted in each treatment group, leading to an artificial safety set of 399 subjects.
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Serious Adverse Events (participants affected / at risk) | 6/133 | 6/133 | 5/133
Other Adverse Events (participants affected / at risk) | 0/133 | 0/133 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab, Pre-filled Syringes (PFS) (N=133) | Canakinumab, Lyophilizate (LYO) (N=133) | Triamcinolone Acetonide (N=133)
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortitis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.